CLINICAL TRIAL: NCT02917421
Title: Accelerated Radiation Therapy (ART) To The Breast And Nodal Stations After Neo-Adjuvant Systemic Therapy And Surgery: A Feasibility Study
Brief Title: Accelerated Radiation Therapy (ART) to the Breast and Nodal Stations
Acronym: ART
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1602017017
Record Dates: First submitted 2016-09-19; First posted 2016-09-28 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1 (Experimental): (Post-segmental Mastectomy, post-mastectomy and Post-mastectomy with expanders or final reconstruction): Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
  Radiation therapy : Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
  Interventions: Radiation: Radiation
- Cohort 2 (Experimental): In addition to receiving radiation to the original tumor bed, patients will also receive radiation to Level III axillary nodes and Supraclavicular nodes: 3D-CRT or IMRT at 2.7 Gy X 15 fraction (40.50 Gy)
  Radiation Therapy : Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — (Post-segmental Mastectomy, post-mastectomy and Post-mastectomy with expanders or final reconstruction): Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.

SUMMARY:
This protocol is for patients with newly diagnosed breast cancer with an indication for post-operative radiotherapy after neo-adjuvant chemotherapy and surgery.

DETAILED DESCRIPTION:
Protocol has two cohorts. Cohort 1 will receive radiation to breast and chest wall. Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy x 15 fractions (40.50 Gy) with a concomitant boost of 0.50 (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.

Cohort 2 patients will receive radiation to breast, chest wall and LevelII/SCV nodes.

In addition to receiving radiation to the original tumor bed, patients will also receive radiation to Level III axillary nodes and Supraclavicular nodes: 3D-CRT or IMRT at 2.7 Gy X 15 fraction (40.50 Gy).

Patients will complete treatment in three weeks (15 fractions). All patients will be followed at 3 months after the completion of treatment then yearly for the next 5 years.

ELIGIBILITY:
The study will also include patients who because of COVID had undergone up to 3 months neoadjuvant hormonal therapy before surgery for clinical T1/T2 BC.

Inclusion Criteria:

* Age older than 18
* Pre- or post-menopausal women with Stage I-III breast cancer
* Status post neoadjuvant systemic therapy
* Status post-chemotherapy breast surgery
* Original biopsy-proven invasive breast cancer, excised with negative margins of at least 1 mm (patients with focally positive margin are not excluded).
* Status post segmental mastectomy or mastectomy, with either negative sentinel node biopsy and/or axillary node dissection (at least 6 nodes removed).
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast and/or nodal area
* Active connective tissue disorders, such as lupus or scleroderma requiring flare therapy
* Pregnant or lactating women
* Concurrent chemotherapy, with the exception of anti HER2neu therapies
* Inadequate axillary dissection in a setting of positive sentinel node
* Patients with more than 5 nodes involved at axillary dissection will be excluded from this study since they will be eligible to receive radiotherapy to level I and II axilla.

Ages: 19 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (3):
- United States (3):
  - New York Presbyterian Hospital - Queens, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: (Post-segmental Mastectomy, post-mastectomy and Post-mastectomy with expanders or final reconstruction): Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
  Radiation therapy : Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
  Radiation: (Post-segmental Mastectomy, post-mastectomy and Post-mastectomy with expanders or final reconstruction):
  Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
- Cohort 2: In addition to receiving radiation to the original tumor bed, patients will also receive radiation to Level III axillary nodes and Supraclavicular nodes: 3D-CRT or IMRT at 2.7 Gy X 15 fraction (40.50 Gy)
  Radiation Therapy : Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
  Radiation: (Post-segmental Mastectomy, post-mastectomy and Post-mastectomy with expanders or final reconstruction):
  Prone whole breast or chest wall 3D-CRT or IMRT at 2.7 Gy X 15 fractions (40.50 Gy) with a concomitant boost of 0.50 Gy (7.5 Gy) to the original tumor bed in post-segmental mastectomy patients or mastectomy scar in post-mastectomy patients. Patients who have undergone reconstruction will not receive concomitant boost.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 47 | 41
Completed | 47 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 47 | 41 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 33 | 62
  >=65 years | 18 | 8 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 39 | 34 | 73
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 10 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 23 | 13 | 36
  More than one race | 12 | 11 | 23
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 41 | 88

OUTCOME MEASURES:

1. Primary Outcome: Acute Toxicity Will be Measured by Evaluating the Number of Patients Who Experience Grade II-III Dermatitis Within 60 Days of Radiation Therapy.
Description: feasibility of accelerated radiotherapy in the post-operative setting of breast cancer patients treated by neo-adjuvant chemotherapy and surgery will be measured, by evaluating the number of patients who experience grade II-III dermatitis within 60 days of the end of treatment. Acute Toxicity will be graded using CTCAE v4.0.
Time Frame: 60 days from start of radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 47 | 41
Participants | 0 | 0

2. Secondary Outcome: Change in Quality of Life of Patients.
Description: The patient reported outcomes or quality of life questionnaires are assessed for the aesthetic and functional outcomes after breast radiation therapy. The score value ranges from 1.00 - 4.00, with a higher score reflecting a poorer outcome. Following is the criteria for evaluating breast radiation therapy outcomes in patients: good (1.00-1.75) ; intermediate (1.76-2.50), fair (2.51 -3.25) and poor (3.26 - 4.00).
Time Frame: Baseline, end of radiation, 1 month post radiation.
Population: Data in the table is representative of those participants who completed the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 46 | 37
score on a scale
  Baseline: number analyzed (Participants) | 45 | 37
  Baseline | 1.62 (0.730) | 1.92 (0.979)
  End of Radiation: number analyzed (Participants) | 46 | 36
  End of Radiation | 1.80 (0.876) | 1.82 (0.855)
  1 month post radiation: number analyzed (Participants) | 37 | 34
  1 month post radiation | 1.59 (0.730) | 1.79 (0.812)

3. Secondary Outcome: Late Radiation Toxicity in Treated Patients
Description: incidence of late radiation toxicity (brachial plexopathy, fibrosis and telangiectasia) will be evaluated and genetic determinants of breast fibrosis will be identified.
Time Frame: 2 years and 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Number of Patients With Grades 2 or Higher Toxicity
Description: Number of patients with grades 2 or higher toxicity
Time Frame: 2 years and 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life of Patients
Description: as for outcome 2
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2025-12

6. Other Pre Specified Outcome: Overall Survival Will be Measured
Time Frame: up to 10 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Molecular Signatures That Predict Fibrosis Will be Prospectively Measured From Blood Samples.
Description: The purpose of this portion of the study will be to collect blood from each subject accrued to the study and willing to donate a specimen of blood for research, to study the TGF-β1 polymorphisms that have been reported to be correlated with the development of fibrosis following radiotherapy for treatment of breast cancer.
Time Frame: 10 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Local Control Rates Will be Measured.
Time Frame: up to 10 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Distant Recurrences Will be Measured.
Time Frame: up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline, 60 days, 2 years and 5 years.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 47/47 | 41/41
Serious Adverse Events (participants affected / at risk) | 2/47 | 0/41
Other Adverse Events (participants affected / at risk) | 45/47 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=47) | Cohort 2 (N=41)
Fever (Infections and infestations) | 1 | 0 — Patient had 100.2 fever (Grade 1, unrelated to the study) with leukopenia and ANC and was COVID positive.
Surgery Wound Infection (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=47) | Cohort 2 (N=41)
Anemia (Blood and lymphatic system disorders) | 3 | 3
Dermatitis, Radiation (Skin and subcutaneous tissue disorders) | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 4 | 10
Lymphedema (Musculoskeletal and connective tissue disorders) | 14 | 9
Fatigue (General disorders) | 21 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Breast Pain (Reproductive system and breast disorders) | 4 | 3
Hot Flashes (Vascular disorders) | 3 | 0
Anxiety (Nervous system disorders) | 3 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 4
Skin Rash (Skin and subcutaneous tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02917421/Prot_SAP_000.pdf